CLINICAL TRIAL: NCT00804258
Title: Integration of Palliative Care in Use of Intra-Peritoneal Chemotherapy for Ovarian Cancer
Brief Title: Palliative Care During Intraperitoneal Chemotherapy in Patients With Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 07007; P30CA033572 (NIH); CHNMC-07007 (Other: NCI PDQ); CDR0000629073 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; stage I ovarian epithelial cancer; stage I ovarian germ cell tumor; stage II ovarian epithelial cancer; stage II ovarian germ cell tumor; stage III ovarian epithelial cancer; stage III ovarian germ cell tumor; stage IV ovarian epithelial cancer; stage IV ovarian germ cell tumor
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Hyperthermic Intraperitoneal Chemotherapy; Early Intervention, Educational; Therapeutics; Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: intraperitoneal chemotherapy
Other: educational intervention
Other: medical chart review
Other: questionnaire administration
Procedure: assessment of therapy complications
Procedure: end-of-life treatment/management
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Palliative care may help improve the quality of life of patients with ovarian cancer who are undergoing intraperitoneal chemotherapy.

PURPOSE: This clinical trial is studying palliative care in patients with ovarian cancer who are undergoing intraperitoneal chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Describe symptoms/concerns before, during, and after intraperitoneal (IP) chemotherapy and the impact of these symptoms/concerns on the quality of life (QOL) of patients with ovarian cancer undergoing IP chemotherapy. (Part I)
* Analyze care received and resource utilization of these patients, including length of hospitalization, ICU admission rates, clinic visits, phone calls, urgent care visits, and other heath system encounters. (Part I)
* Develop palliative care assessment measures and interventions that apply to IP chemotherapy. (Part II)
* Implement a palliative care intervention in a pilot of 6 patients. (Part II)
* Describe the impact of implementing palliative care interventions on resource utilization, improved QOL and symptoms, and number of chemotherapy courses completed. (Part II)

OUTLINE: This is a two-part study.

* Part I (retrospective portion): Patients who have undergone intraperitoneal (IP) chemotherapy within the past 6-12 months undergo a retrospective interview and chart audit to identify their needs and experiences.
* Part I (prospective portion): Patients are followed monthly for up to 6 months during IP chemotherapy to provide information about usual care and to identify needs and palliative care concerns. Patients also complete a quality-of-life (QOL) questionnaire (COH QOL Ovarian tool) and undergo a prospective interview.
* Part II (intervention): Patients undergo comprehensive palliative care assessment, a patient teaching session prior to the initiation of IP chemotherapy, and a palliative care intervention during IP chemotherapy. Patients also complete a QOL questionnaire and undergo an interview. Patients are followed monthly for up to 6 months during IP chemotherapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of ovarian cancer
* Under the care of the Medical Oncology Department at the City of Hope National Medical Center
* Undergoing intraperitoneal chemotherapy

PATIENT CHARACTERISTICS:

* Life expectancy > 6 months
* Speaks English or Spanish

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under the care of the Medical Oncology department at the City of Hope
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2007-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Symptoms/concerns before, during, and after intraperitoneal (IP) chemotherapy and their impact on quality of life (QOL) | 6 months from study entry
Length of hospitalization, ICU admission rates, clinic visits, phone calls, urgent care visits, and other heath system encounters | 6 months from study entry
Development of palliative care assessment measures and interventions that apply to IP chemotherapy | 6 months from study start
Implementation of a palliative care intervention | 6 months from study entry
Impact of implementing palliative care interventions on resource utilization, improved QOL and symptoms, and number of chemotherapy courses completed | 6 months from study entry

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Grant, RN, DNSc, FAAN, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States